CLINICAL TRIAL: NCT06589661
Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' Experience During and After Unexpected Cesarean Delivery Under General Anesthesia to Inform Anesthetic Practice. A Prospective Patient-centred Multidisciplinary Mixed-method. (PAS-EDU-uCD-GA)
Brief Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' Experience During and After Unexpected Cesarean Delivery Under General Anesthesia to Inform Anesthetic Practice
Acronym: PAS-EDU-uCD-GA
Status: Recruiting | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24-07
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Psychological Well Being
Keywords: cesarean delivery; patient experience; general anesthetic
MeSH Terms: conditions — Psychological Well-Being | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unexpected cesarean delivery under general anesthesia: Patients who have an unexpected cesarean delivery under general anesthesia.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patients will be interviewed by the research team to learn about their experience of Cesarean delivery under general anesthetic.

SUMMARY:
This study aims to explore the patients' and providers' perspectives and inform future anesthetic practice for patients undergoing unexpected cesarean delivery (CD) under general anesthetic (GA). The consideration of patients' concerns, preferences, expectations, and suggestions may lead to enhanced patient satisfaction, compliance, and quality of care that future patients receive during unexpected CD under GA. The investigators will possibly be able to identify gaps in procedural performance that warrant further investigation during the second phase of this study which will contribute to improvement of overall patient care. During the third phase, educational material will be generated from patient insights and will be distributed to the Department of Anesthesia, Department of Obstetrics and Gynaecology, Labour and Delivery Nurses and team of Anesthesia Assistants and Respiratory Therapists.

DETAILED DESCRIPTION:
Cesarean delivery (CD) is a surgical procedure that allows for birth of a neonate through a laparotomy and hysterotomy and is the most common surgical procedure performed worldwide with 21% of all childbirths occurring via CD.

A single-shot spinal anesthesia is the most common technique for CD due to its simplicity, quality of sensory blockade and reliability, as well as because of the safety for the fetus. Nevertheless, there are clinical situation where general anesthesia is necessary. General anesthesia care in obstetric scenarios remains a serious concern because of a high failed intubation rate, accidental awareness, increasing association with postpartum depression requiring hospitalization, suicidal ideation and self-inflicted injury, and traumatic birth experiences. General anesthesia for CD might not be planned and pivoting to this unexpected type of anesthesia can be a traumatic experience for patients and their families. Patients may receive a GA for various reasons, including failed neuraxial anesthesia, hemodynamic instability, or critical fetal situations not amendable to neuraxial anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* English language proficiency (as interviews will be performed in English)
* ASA Physical Classification Score 2-5 +/- E
* Emergency or Urgent Cesarean Delivery with the need for general anesthesia due to fetal or maternal emergencies (e.g., fetal bradycardia, HELLP syndrome, etc.)
* Unexpected Cesarean Delivery is defined as Level 1 (Emergency - Immediate threat to life of woman or fetus) and Level 2 (Urgent - Maternal or fetal compromise which is not immediately life-threatening) Cesarean Deliveries.21
* Patients will be included if they undergo preterm delivery (under 37 weeks of gestation, or are having a multiple gestation pregnancy, also, if there is a significant fetal anomaly present.

Exclusion criteria:

* Under 18 years of age
* Unable to answer questions due to a language barrier or because of their mental or physical state (e.g., intubated patients)
* BMI at the time of delivery that falls in the super-morbidly obese category (BMI > 55 kg/m2)
* Patients who underwent preterm delivery (under 32 weeks gestation)
* Patients will be excluded if neonatal death has occurred.
* Patients who were scheduled for an elective Cesarean Delivery, but had contraindicated or failed neuraxial anesthesia and required general anesthesia for or during their CD will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who deliver by unexpected cesarean section under general anesthesia at Mount Sinai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | Following cesarean delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be asked to rate their experience of having a cesarean delivery under general anesthesia, in terms of satisfaction and their experience with any discomfort. Some questions are yes/no, some are on a scale from 1-10, where 1 = not at all and 10 = totally agree, and some are open-ended. The questionnaire will take approximately 10 minutes to complete.
Patient interview | Following cesarean delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be interviewed in person by a member of the research team and asked open ended questions. Interviews will be recorded, transcribed and coded for themes. Responses are not reported on any scale. The interview will take approximately 30 minutes to complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No